CLINICAL TRIAL: NCT01850914
Title: Vascular Risk Factors, Subclinical and Manifest Vascular Disease in Patients With Idiopathic Normal Pressure Hydrocephalus
Brief Title: Vascular Risk Factors in INPH-patients
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Hanna Israelsson, MD, PhD-student, Umeå University
Other Study IDs: 2011-52-31M; Dnr 2011-52-31M (Other: Regional Ethics Board in Umeå)
Record Dates: First submitted 2013-04-04; First posted 2013-05-10 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Hydrocephalus, Normal Pressure; Vascular Diseases; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases
Keywords: Normal pressure hydrocephalus; Vascular risk factors
MeSH Terms: conditions — Hydrocephalus, Normal Pressure; Vascular Diseases; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Shunted patients with INPH: Cases: Patients with normal pressure hydrocephalus who have underwent surgery. Controls: Sex- and age-matched community based controls.
- Populationbased elderly.: A group of populationbased elderly, matched according to age and sex to the patients with INPH. Vascular risk factors studied.

SUMMARY:
Idiopathic normal pressure hydrocephalus (INPH) is a treatable and a common disease of the elderly. The overall objective of this work is to describe cardio- and cerebrovascular risk factors and vascular disease in shunted INPH-patients compared to an age- and sex matched elderly population, as well as the impact of vascular risk factors and vascular co-morbidity on clinical symptoms and outcome of surgery in INPH-patients. The hypothesis is that INPH-patients have a higher level of vascular risk factors and subclinical organ damage than a normal elderly population, and that the higher the level of existing vascular risk factors, the more severe the symptoms of the hydrocephalic disease.

ELIGIBILITY:
Inclusion Criteria:

* INPH-patients who underwent surgery 2008-2010 and registered in the Swedish National Register of Hydrocephalus
* age <60 and >85
* (only for controls) living in Umeå

Exclusion Criteria:

* death
* a known mini mental state estimation <23
* inability to communicate (because of severe stroke, aphasia, dementia)
* (only for controls) individuals with INPH who has not yet underwent surgery, or has not been chosen to undergo surgery.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases are all INPH-patients who underwent surgery 2008-2010 and are registered in the Swedish National Register of Hydrocephalus. Controls were found in the Swedish population indox of Umeå, and were indivdually matched to cases according to age and sex.
Sampling Method: Probability Sample
Enrollment: 860 (Actual)
Dates: Start 2010-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Differences in bloodpressure between INPH-patients and a sex- and agematched community based population | More than two weeks, not longer than 6 months.
  Enrollment of participants 2010-2012. First, all participants complete a questionnaire, second they go to their local health care center or nearby hospital for measurements and blood samples. The visit at the health care center/hospital is within a couple of months. Participants are not followed further (cross-sectional study). Analyses performed 2013-2014. First results approximately reported in the end of 2013.

SECONDARY OUTCOMES:
Quality of Life in INPH-patients compared to a sex- and age-matched population. | More than 2 weeks, not longer than 6 months.
  Enrollment of participants 2010-2012. First, all participants complete a questionnaire, second they go to their local health care center or nearby hospital for measurements and blood samples. The visit at the health care center/hospital is within a couple of months. Participants are not followed further (cross-sectional study). Analyses performed 2013-2014. First results approximately reported in the end of 2013.

OTHER OUTCOMES:
Differences between INPH-patients and community based controls regarding smoking. | More than two weeks, not longer than 6 months.
  Enrollment of participants 2010-2012. First, all participants complete a questionnaire, second they go to their local health care center or nearby hospital for measurements and blood samples. The visit at the health care center/hospital is within a couple of months. Participants are not followed further (cross-sectional study). Analyses performed 2013-2014. First results approximately reported in the end of 2013.
Differences between INPH-patients and community based controls regarding waist-to-hip ratio. | More than 2 weeks, not longer than 6 months.
  Enrollment of participants 2010-2012. First, all participants complete a questionnaire, second they go to their local health care center or nearby hospital for measurements and blood samples. The visit at the health care center/hospital is within a couple of months. Participants are not followed further (cross-sectional study). Analyses performed 2013-2014. First results approximately reported in the end of 2013.
Differences between INPH-patients and community based controls regarding dietary risk score. | More than 2 weeks, not more than 6 months.
  Enrollment of participants 2010-2012. First, all participants complete a questionnaire, second they go to their local health care center or nearby hospital for measurements and blood samples. The visit at the health care center/hospital is within a couple of months. Participants are not followed further (cross-sectional study). Analyses performed 2013-2014. First results approximately reported in the end of 2013.
Differences between INPH-patients and community based controls regarding physical activity. | More than 2 weeks, not longer than 6 months.
  Enrollment of participants 2010-2012. First, all participants complete a questionnaire, second they go to their local health care center or nearby hospital for measurements and blood samples. The visit at the health care center/hospital is within a couple of months. Participants are not followed further (cross-sectional study). Analyses performed 2013-2014. First results approximately reported in the end of 2013.
Differences between INPH-patients and community based controls regarding diabetes mellitus. | More than 2 weeks, not longer than 6 months.
  Enrollment of participants 2010-2012. First, all participants complete a questionnaire, second they go to their local health care center or nearby hospital for measurements and blood samples. The visit at the health care center/hospital is within a couple of months. Participants are not followed further (cross-sectional study). Analyses performed 2013-2014. First results approximately reported in the end of 2013.
Differences between INPH-patients and community based controls regarding alcohol intake. | More than 2 weeks, not longer than 6 months.
  Enrollment of participants 2010-2012. First, all participants complete a questionnaire, second they go to their local health care center or nearby hospital for measurements and blood samples. The visit at the health care center/hospital is within a couple of months. Participants are not followed further (cross-sectional study). Analyses performed 2013-2014. First results approximately reported in the end of 2013.
Differences between INPH-patients and community based controls regarding psychosocial factors. | More than 2 weeks, not longer than 6 months.
  Enrollment of participants 2010-2012. First, all participants complete a questionnaire, second they go to their local health care center or nearby hospital for measurements and blood samples. The visit at the health care center/hospital is within a couple of months. Participants are not followed further (cross-sectional study). Analyses performed 2013-2014. First results approximately reported in the end of 2013.
Differences between INPH-patients and community based controls regarding cardiac causes. | More than two weeks, not longer than 6 weeks.
  Enrollment of participants 2010-2012. First, all participants complete a questionnaire, second they go to their local health care center or nearby hospital for measurements and blood samples. The visit at the health care center/hospital is within a couple of months. Participants are not followed further (cross-sectional study). Analyses performed 2013-2014. First results approximately reported in the end of 2013.
Differences between INPH-patients and community based controls regarding ratio of apolipoprotein B to A1. | More than 2 weeks, not longer than 6 months.
  Enrollment of participants 2010-2012. First, all participants complete a questionnaire, second they go to their local health care center or nearby hospital for measurements and blood samples. The visit at the health care center/hospital is within a couple of months. Participants are not followed further (cross-sectional study). Analyses performed 2013-2014. First results approximately reported in the end of 2013.
Differences between INPH-patients and community based controls regarding activities of daily life (ADL). | More than 2 weeks, not longer than 6 months.
  Enrollment of participants 2010-2012. First, all participants complete a questionnaire, second they go to their local health care center or nearby hospital for measurements and blood samples. The visit at the health care center/hospital is within a couple of months. Participants are not followed further (cross-sectional study). Analyses performed 2013-2014. First results approximately reported in the end of 2013.
Differences between INPH-patients and community based controls regarding frequency, severity and fear of falling. | More than 2 weeks, not longer than 6 months.
  Enrollment of participants 2010-2012. First, all participants complete a questionnaire, second they go to their local health care center or nearby hospital for measurements and blood samples. The visit at the health care center/hospital is within a couple of months. Participants are not followed further (cross-sectional study). Analyses performed 2013-2014. First results approximately reported in the end of 2013.
Differences between INPH-patients and community based controls regarding headache. | More than2 weeks, not longer than 6 months.
  Enrollment of participants 2010-2012. First, all participants complete a questionnaire, second they go to their local health care center or nearby hospital for measurements and blood samples. The visit at the health care center/hospital is within a couple of months. Participants are not followed further (cross-sectional study). Analyses performed 2013-2014. First results approximately reported in the end of 2013.
Differences between INPH-patients and community based controls regarding epilepsy. | More than 2 weeks, not longer than 6 months.
  Enrollment of participants 2010-2012. First, all participants complete a questionnaire, second they go to their local health care center or nearby hospital for measurements and blood samples. The visit at the health care center/hospital is within a couple of months. Participants are not followed further (cross-sectional study). Analyses performed 2013-2014. First results approximately reported in the end of 2013.
Differences between INPH-patients and community based controls regarding kidney function. | More than 2 weeks, not longer than 6 months.
  Enrollment of participants 2010-2012. First, all participants complete a questionnaire, second they go to their local health care center or nearby hospital for measurements and blood samples. The visit at the health care center/hospital is within a couple of months. Participants are not followed further (cross-sectional study). Analyses performed 2013-2014. First results approximately reported in the end of 2013.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Malm, MD, PhD, Study Director — Umeå University, Departement of Pharmacology and Clinical Neuroscience; Hanna Israelsson, MD, PhD-stud, Principal Investigator — Umeå University, Departement of Pharmacology and Clinical Neuroscience
Locations (1):
- Umeå University, Umeå University Hospital, Departement of Pharmacology and Clinical Neuroscience, Umeå, Västerbotten County, Sweden

REFERENCES:
- [Derived] Eklund SA, Israelsson H, Carlberg B, Malm J. Vascular risk profiles for predicting outcome and long-term mortality in patients with idiopathic normal pressure hydrocephalus: comparison of clinical decision support tools. J Neurosurg. 2022 Jun 10;138(2):476-482. doi: 10.3171/2022.4.JNS22125. Print 2023 Feb 1. PMID 35901765